CLINICAL TRIAL: NCT05147779
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cells for the Treatment of Peyronie's Disease, Erectile Dysfunction, and Interstitial Cystitis
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Stem Cells for Peyronie's Disease, ED, and Interstitial Cystitis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-1-MSC-015
Record Dates: First submitted 2021-11-29; First posted 2021-12-07 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Erectile Dysfunction; Peyronie's Disease; Interstitial Cystitis
Keywords: Erectile Dysfunction; Peyronie's Disease; stem cell treatment; Interstitial Cystitis
MeSH Terms: conditions — Erectile Dysfunction; Penile Induration; Cystitis, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (AlloRx) (Experimental): intravenous and intracavernosal or interstitial delivery (total dose of 100 million cells)
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous and intracavernosal or interstitial delivery of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of Peyronie's disease, erectile dysfunction , and Interstitial Cystitis

DETAILED DESCRIPTION:
This patient funded trial aims to study the safety and efficacy of intravenous and intracavernosal or interstitial delivery of cultured allogeneic adult umbilical cord derived mesenchymal stem cells (UC-MSCs) for the treatment of Peyronie's disease, erectile dysfunction , and Interstitial Cystitis. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Peyronie's Disease, erectile dysfunction, or Interstitial Cystitis
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (1):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Demour S, Jafar H, Adwan S, AlSharif A, Alhawari H, Alrabadi A, Zayed A, Jaradat A, Awidi A. Safety and Potential Therapeutic Effect of Two Intracavernous Autologous Bone Marrow Derived Mesenchymal Stem Cells injections in Diabetic Patients with Erectile Dysfunction: An Open Label Phase I Clinical Trial. Urol Int. 2018;101(3):358-365. doi: 10.1159/000492120. Epub 2018 Aug 31. PMID 30173210
- [Background] Bahk JY, Jung JH, Han H, Min SK, Lee YS. Treatment of diabetic impotence with umbilical cord blood stem cell intracavernosal transplant: preliminary report of 7 cases. Exp Clin Transplant. 2010 Jun;8(2):150-60. PMID 20565373
- [Background] Levy JA, Marchand M, Iorio L, Zribi G, Zahalsky MP. Effects of Stem Cell Treatment in Human Patients With Peyronie Disease. J Am Osteopath Assoc. 2015 Oct;115(10):e8-13. doi: 10.7556/jaoa.2015.124. PMID 26414724